CLINICAL TRIAL: NCT05909163
Title: Spoken Language Biomarker of Cognitive Impairment in PD
Brief Title: Spoken Discourse Biomarker of PD Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Angela Roberts, Principal Investigator, Northwestern University
Other Study IDs: STU00209602
Record Dates: First submitted 2021-10-21; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pakinson's disease without cognitive impairment: * Age 50-90 years
  * Diagnosis of idiopathic Parkinson's disease (UK Brain Bank criteria) made by a movement disorders specialist
  * Under the care of a movement disorders specialist for a minimum of 1-year duration
  * Native monolingual English speaker
  * Hoehn & Yahr score between 1.5 and 4
  * Grade 10 education, or higher
  * Sufficient vision and hearing (aided or unaided) for all experiment tasks
  * Montreal Cognitive Assessment (or MoCA-converted MMSE score) greater than or equal to 25
  * No subjective complaints of cognitive difficulty or word finding issues
- Pakinson's disease with cognitive impairment: * Age 50-90 years
  * Diagnosis of idiopathic Parkinson's disease (UK Brain Bank criteria) made by a movement disorders specialist
  * Under the care of a movement disorders specialist for a minimum of 1-year duration
  * Native monolingual English speaker
  * Hoehn & Yahr score between 1.5 and 4
  * Grade 10 education, or higher
  * Sufficient vision and hearing (aided or unaided) for all experiment tasks
  * Montreal Cognitive Assessment (or MoCA-converted MMSE score) greater than or equal to 17
  * Subjective complaints of cognitive difficulty or word finding issues, without significant impact on activities of daily living

SUMMARY:
The purpose of this study is to identify unique profiles of speech and language changes that distinguish individuals with Parkinson's disease from adults without Parkinson's disease and individuals with Parkinson's disease with cognitive (e.g., memory, thinking skills) impairment from those without cognitive impairment.

DETAILED DESCRIPTION:
Aim 1 will characterize PD-MCI (Parkinson's disease mild cognitive impairment), PDN (Parkinson's disease without cognitive impairment), and HA (healthy adult) spoken discourse, cognitive, and motor speech profiles. Phase 2 biomarker development requires robustly characterized cohorts in which to test candidate biomarkers. Using a standardized battery of cognitive, language, and motor speech tests PD participants will be assigned to PD-MCI (single/multi-domain) or PDN groups. The investigators propose collecting spoken discourse samples using standardized elicitation protocols. The same tasks will be extracted from the extant HA database. Researchers will transcribe, code, and analyze discourse samples. Group differences (including sub-analyses for single and multi-domain MCI subtypes), elicitation stimuli effects, and group x stimuli interactions will be examined using multivariate and mixed-design ANOVA procedures.

Aim 2 will develop and evaluate the classification accuracy of an optimally weighted discourse classification function for PD-MCI and PDN. The investigators propose using discriminant function analysis to identify an optimized composite variable that best predicts PD-MCI, PDN, and HA group membership. Sensitivity/specificity analyses, positive/negative predictive values, and receiver operating characteristic curves will be used to evaluate the discourse classification function properties.

The primary endpoint is an optimally weighted discourse function that can classify PD-MCI with > 80% sensitivity/specificity.

ELIGIBILITY:
Inclusion Criteria:

Only individuals with PD will be newly recruited and enrolled as part of the study. Healthy adult data will be extracted from extant databases (publicly available) from NIH-funded studies.

Inclusion Criteria Person with Parkinson's disease without cognitive impairment

* Age 50-90 years
* Diagnosis of idiopathic Parkinson's disease (UK Brain Bank criteria) made by a movement disorders specialist
* Under the care of a movement disorders specialist for a minimum of 1-year duration
* Native monolingual English speaker
* Hoehn & Yahr score between 1.5 and 4
* Grade 10 education, or higher
* Sufficient vision and hearing (aided or unaided) for all experiment tasks
* Montreal Cognitive Assessment (or MoCA-converted MMSE score) greater than or equal to 25
* No subjective complaints of cognitive difficulty or word finding issues

Inclusion Criteria Person with Parkinson's disease mild cognitive impairment

* Age 50-90 years
* Diagnosis of idiopathic Parkinson's disease (UK Brain Bank criteria) made by a movement disorders specialist
* Under the care of a movement disorders specialist for a minimum of 1-year duration
* Native monolingual English speaker
* Hoehn & Yahr score between 1.5 and 4
* Grade 10 education, or higher
* Sufficient vision and hearing (aided or unaided) for all experiment tasks
* Montreal Cognitive Assessment (or MoCA-converted MMSE score) greater than or equal to 17
* Subjective complaints of cognitive difficulty or word finding issues, without significant impact on activities of daily living

Inclusion Healthy Adults (from extant data base - no new recruiting)

* Age 50-90 years
* Montreal Cognitive Assessment (or MoCA-converted MMSE score) greater than or equal to 26
* Native monolingual English speaker
* Grade 10 education, or higher
* Sufficient vision and hearing (aided or unaided) for all experiment tasks

Exclusion Criteria:

Exclusion Criteria Neurological injury or disease (other than PD for the PD cohort)

* History of unmanaged or untreated depression or major psychiatric illness
* History of deep brain stimulation surgery (DBS)
* Diagnosis of Dementia with Lewy Bodies

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only individuals with PD will be newly recruited and enrolled as part of the study. Healthy adult data will be extracted from extant databases (publicly available) from NIH-funded studies.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Discourse Composite Variable | baseline
  Weighted variable comprised of discourse features extracted from spoken discourse samples across productivity, lexical retrieval, verbal fluency, syntax complexity, grammatical accuracy, narrative coherence, correct information units, and main event accuracy. Raw data from each measure are multiplied by a specified weight and summed to generate a single composite discourse score.

SECONDARY OUTCOMES:
Words per minute | baseline
  Number of total words ÷ Participant speaking time in minutes
Correct information units (CIUs) | baseline
  Number of words intelligible in context and accurate, relevant, and informative about the picture content (Brookshire & Nicholas, 1994; Nicholas & Brookshire, 1993)
% CIUs | baseline
  CIUs ÷ number of words (Brookshire & Nicholas, 1994; Nicholas & Brookshire, 1993) × 100
CIUs/min | baseline
  CIUs ÷ Participant speaking time in minutes (Brookshire & Nicholas, 1994; Nicholas & Brookshire, 1993)
% Main Events | baseline
  Proportion of correct narrative main events (Capilouto et al., 2005)
Moving-average type-token ratio (MATTR) | baseline
  SALT-generated moving-average ratio of different words : total words (SALT Inc., 2017"). Window size = 23 words, based on the number of words in smallest discourse sample (Roberts & Post, 2018)
Mean length of utterance (MLU) | baseline
  Mean length of utterance in words for intelligible, complete, verbal, task-relevant utterances (SALT Inc., 2017)
% Grammatical | baseline
  Number of content units without lexical selection or grammar rule violations (Thompson et al., 1995, 2012) ÷ Total intelligible, complete, verbal, task-relevant utterances × 100
Subordination index (SI) | baseline
  Subordination index composite score. The ratio of total number of subject + Predicate clauses : total number of content units (SALT Software LLC, 2018b)
Number of clauses/content units | baseline
  Number of clauses per content units (based on the count of main verbs)
Word-level dysfluencies/content units | baseline
  Total number of word, syllable, and sound repetitions plus the total number of initial, middle, and final sound prolongations (SALT Software LLC, 2018a) ÷ Total utterances
Number of pauses/content units | baseline
  Number of pauses >1.5 s ÷ Total utterances
Percent maze words/total words | baseline
  Maze words (i.e., filled pauses, false starts, reformulations, and interjections) ÷ Maze words + non-maze words

OTHER OUTCOMES:
Discourse Global Coherence | baseline
  Each utterance is rated on a scale of 1-4 judging the relation of each sentence to the overall topic. '4' reflects that the utterance is overtly related to the stimulus as defined by mention of actors, actions, and/or objects present in the stimulus, which are of significant importance to the main details of the stimulus.
Discourse Local Coherence | baseline
  Each utterance is rated on a scale of 1-5 judging the relation of adjacent sentences to each other. '5' reflects that the utterance is in relation to continuation, elaboration, repetition, subordination or coordination of ideas from the preceding utterance.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Evanston, Illinois, United States

REFERENCES:
- [Background] Nicholas LE, Brookshire RH. A system for quantifying the informativeness and efficiency of the connected speech of adults with aphasia. J Speech Hear Res. 1993 Apr;36(2):338-50. doi: 10.1044/jshr.3602.338. PMID 8487525
- [Background] Brookshire RH, Nicholas LE. Speech sample size and test-retest stability of connected speech measures for adults with aphasia. J Speech Hear Res. 1994 Apr;37(2):399-407. doi: 10.1044/jshr.3702.399. PMID 8028321
- [Background] Capilouto G, Wright HH, Wagovich SA. CIU and main event analyses of the structured discourse of older and younger adults. J Commun Disord. 2005 Nov-Dec;38(6):431-44. doi: 10.1016/j.jcomdis.2005.03.005. Epub 2005 Apr 26. PMID 16199238
- [Background] Roberts A, Post D. Information Content and Efficiency in the Spoken Discourse of Individuals With Parkinson's Disease. J Speech Lang Hear Res. 2018 Sep 19;61(9):2259-2274. doi: 10.1044/2018_JSLHR-L-17-0338. PMID 30208482
- [Background] Thompson CK, Cho S, Hsu CJ, Wieneke C, Rademaker A, Weitner BB, Mesulam MM, Weintraub S. Dissociations Between Fluency And Agrammatism In Primary Progressive Aphasia. Aphasiology. 2012;26(1):20-43. doi: 10.1080/02687038.2011.584691. PMID 22199417
- [Background] Thompson, C. K., Shapiro, L. P., Li, L., & Schendel, L. (1995). Analysis of verbs and verb-argument structure: A method for quantification of aphasic language production. Clinical Aphasiology, 23, 121-140.
- [Background] Harris Wright, H., Koutsoftas, A., Fergadiotis, G., & Capilouto, G. (2010). Coherence in Stories Told by Adults With Aphasia.
- [Background] Wright HH, Capilouto GJ. Considering a multi-level approach to understanding maintenance of global coherence in adults with aphasia. Aphasiology. 2012 Jan 1;26(5):656-672. doi: 10.1080/02687038.2012.676855. Epub 2012 May 10. PMID 22962509
- [Background] Glosser G, Deser T. Patterns of discourse production among neurological patients with fluent language disorders. Brain Lang. 1991 Jan;40(1):67-88. doi: 10.1016/0093-934x(91)90117-j. PMID 2009448
- [Background] Van Leer E, Turkstra L. The effect of elicitation task on discourse coherence and cohesion in adolescents with brain injury. J Commun Disord. 1999 Sep-Oct;32(5):327-48; quiz 348-9. doi: 10.1016/s0021-9924(99)00008-8. PMID 10498013
- See also: SALT Subordination index — https://www.saltsoftware.com/media/wysiwyg/codeaids/SI_Scoring_Guide.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT05909163/Prot_SAP_000.pdf